CLINICAL TRIAL: NCT04434066
Title: A Comparison of Perioperative and Patient-Centered Outcomes with Abdominal Versus Vaginal Morcellation: a Randomized-Controlled Trial
Brief Title: Outcomes on Abdominal Versus Vaginal Morcellation At Time of Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kimberly Kho, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-1402
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Abnormal Uterine Bleeding; Uterine Bleeding; Fibroid Uterus; Surgery
Keywords: hysterectomy; abnormal uterine bleeding; morcellation; abdominal; vaginal; surgery; laparoscopic; laparoscopy; total hysterectomy; pelvic pain; endometriosis
MeSH Terms: conditions — Metrorrhagia; Uterine Hemorrhage; Leiomyoma; Pelvic Pain; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abdominal Morcellation (Experimental): Abdominal morcellation will occur following completion of the hysterectomy. Route of incision will be either suprapubic or umbilical incision - based on surgeon preferences. All steps and instruments have been standardized for abdominal morcellation.
  Interventions: Procedure: Total Laparoscopic Hysterectomy
- Vaginal Morcellation (Experimental): Vaginal morcellation will occur following completion of the hysterectomy. All steps and instruments have been standardized for vaginal morcellation.
  Interventions: Procedure: Total Laparoscopic Hysterectomy

INTERVENTIONS:
Procedure: Total Laparoscopic Hysterectomy — Participants will be randomized into either abdominal or vaginal morcellation at time of total laparoscopic hysterectomy

SUMMARY:
The purpose of the study is to investigate differences in perioperative and postoperative outcomes between the abdominal (AM) versus vaginal (VM) routes of contained morcellation in participants undergoing laparoscopic total hysterectomies in a randomized controlled trial.

DETAILED DESCRIPTION:
The purpose of the proposed study is to investigate differences in intraoperative and postoperative outcomes between the abdominal (AM) versus vaginal (VM) routes of contained morcellation in subjects undergoing laparoscopic total hysterectomies in a randomized surgical trial.

Objectives:

1. To evaluate differences in total operating time between subjects undergoing AM compared to VM.
2. To evaluate differences in morcellation time between AM and VM.
3. To evaluate differences in the amount of total narcotic use during hospital admission between AM and VM through morphine milligram equivalents (MME).
4. To evaluate differences in the patient's subjective pain assessment via Visual Analogue Scale (VAS) before surgery, at 2-weeks, and at 6 week post-operative visits in both AM and VM groups.
5. To evaluate differences in the patient's pain medication usage as reported by the patient verbally at 24-hours post-operatively and 2-weeks post surgery between AM and VM groups.
6. To evaluate differences in body image survey (BIS) scores at enrollment and 6-week postoperative visit between the AM group compared to VM group.
7. To evaluate differences in overall Quality of Life (QoL) scores at enrollment and 6-week postoperative visit between the AM group compared to VM group.
8. To evaluate differences in Quality of Recovery (QoR) scores at enrollment and at 24-hours post-operatively, and then 2-weeks post surgery between AM and VM group.

ELIGIBILITY:
Inclusion Criteria:

* All benign total laparoscopic hysterectomy and/or robotic-assisted hysterectomy, +/- unilateral salpingo-oophorectomy or bilateral salpingo-oophorectomy
* Adnexectomy, cystectomy, tubal procedures at time of hysterectomy
* Age >18 years old
* Uterus >12 weeks, or >250 grams (based on imaging), or requiring morcellation based on clinical judgment at time of pre-operative enrollment
* English and Spanish speaking

Exclusion Criteria:

* Pre-malignant conditions (i.e. endometrial intraepithelial neoplasia, high-grade cervical intraepithelial neoplasia), known gynecologic malignancy, and any contraindications to abdominal or vaginal morcellation
* Planned concurrent procedures (i.e. hernia repair, bowel resections, anti-incontinence procedures, prolapse repair, and mastectomy)
* Appendectomy for endometriosis is not excluded
* No chronic pain disorders requiring medical management (endometriosis can be included)
* Planned abdominal hysterectomy or vaginal hysterectomy candidates
* Conversion to laparotomy or inability to complete morcellation
* Contraindications to laparoscopy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All females
Enrollment: 46 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Mean difference in total operating room time | intraoperative
  Total operating room time is defined as skin incision to skin closure

SECONDARY OUTCOMES:
Mean difference from baseline in Body Image Scale Score to 6-weeks post-operatively | through study completion up to 6-weeks post-operatively
  Body Image Scale will be collected at baseline, and 6-weeks post-operatively. Body Image Scale will be scored from 10 to 40 points maximum, with higher scores referring to being "very dissatisfied" with overall body image
Mean difference from baseline in Pain Visual Analogue Scale to 6-weeks post-operatively | through study completion up to 6-weeks post-operatively
  Pain Visual Analogue Scale will be collected at baseline, and 6-weeks post-operatively. VAS scale will be measured from 0 to 10mm, with higher scores referring to more pain experienced
Mean difference from baseline in Quality of Recovery Score to 2-weeks post-operatively | through study completion up to 6-weeks post-operatively
  Quality of Recovery will be collected at baseline, 24-hours, and 2-weeks post-operatively. Quality of Recovery will be scored from 10 to 100, with higher scores referring to better quality of recovery
Mean difference from baseline in Quality of Life Score to 6-weeks post-operatively | through study completion up to 6-weeks post-operatively
  Quality of Life Scores will be collected at baseline, and 6-weeks post-operatively. The Quality of Life Score will be scored from 11 to 44, with higher scores referring to better quality of life
Morcellation Time | intraoperative
  Defined as specimen bag introduction to specimen bag removal
Rates of Post-Operative Complications | through study completion up to 6-weeks post-operatively
  Post-operative complications will be collected including: readmission to the hospital or emergency room, number of visits seen in the clinic, diagnoses of infection, bleeding, blood transfusions, surgery-related injuries, reoperations, and overall mortality
Mean difference in the dosages of morphine milligram equivalent (MME) for post-operative pain between abdominal and vaginal morcellation | after surgery to 2-weeks post-operatively
  The type and dosages of various narcotics will be recorded between both groups following surgery until 2-weeks post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Kho, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] US Food and Drug Administration. Laparoscopic Uterine Power Morcellation in Hysterectomy and Myomectomy. US FDA, Silver Spring, MD; 2014 (FDA Safety Communication)
- [Background] US Food and Drug Administration. Updated Laparoscopic Uterine Power Morcellation in Hysterectomy and Myomectomy. US FDA, Silver Spring, MD; 2014 (FDA Safety Communication)
- [Background] Siedhoff MT, Cohen SL. Tissue Extraction Techniques for Leiomyomas and Uteri During Minimally Invasive Surgery. Obstet Gynecol. 2017 Dec;130(6):1251-1260. doi: 10.1097/AOG.0000000000002334. PMID 29112659
- [Background] Cohen SL, Einarsson JI, Wang KC, Brown D, Boruta D, Scheib SA, Fader AN, Shibley T. Contained power morcellation within an insufflated isolation bag. Obstet Gynecol. 2014 Sep;124(3):491-497. doi: 10.1097/AOG.0000000000000421. PMID 25162248
- [Background] Solima E, Scagnelli G, Austoni V, Natale A, Bertulessi C, Busacca M, Vignali M. Vaginal Uterine Morcellation Within a Specimen Containment System: A Study of Bag Integrity. J Minim Invasive Gynecol. 2015 Nov-Dec;22(7):1244-6. doi: 10.1016/j.jmig.2015.07.007. Epub 2015 Jul 20. PMID 26205578
- [Background] Moawad GN, Abi KhalIL ED, Opoku-Anane J, Marfori CQ, Harman AC, Fisher S, Levy M, Robinson JK. Comparison of methods of morcellation: manual versus power. Acta Obstet Gynecol Scand. 2016 Jan;95(1):52-4. doi: 10.1111/aogs.12783. Epub 2015 Oct 19. PMID 26400045
- [Background] Meurs EAIM, Brito LG, Ajao MO, Goggins ER, Vitonis AF, Einarsson JI, Cohen SL. Comparison of Morcellation Techniques at the Time of Laparoscopic Hysterectomy and Myomectomy. J Minim Invasive Gynecol. 2017 Jul-Aug;24(5):843-849. doi: 10.1016/j.jmig.2017.04.023. Epub 2017 May 5. PMID 28483536
- [Background] Venturella R, Rocca ML, Lico D, La Ferrera N, Cirillo R, Gizzo S, Morelli M, Zupi E, Zullo F. In-bag manual versus uncontained power morcellation for laparoscopic myomectomy: randomized controlled trial. Fertil Steril. 2016 May;105(5):1369-1376. doi: 10.1016/j.fertnstert.2015.12.133. Epub 2016 Jan 19. PMID 26801067
- [Background] Frasca C, Degli Esposti E, Arena A, Tuzzato G, Moro E, Martelli V, Seracchioli R. Can In-Bag Manual Morcellation Represent an Alternative to Uncontained Power Morcellation in Laparoscopic Myomectomy? A Randomized Controlled Trial. Gynecol Obstet Invest. 2018;83(1):52-56. doi: 10.1159/000477171. Epub 2017 Jun 7. PMID 28586771
- [Background] Ghezzi F, Cromi A, Uccella S, Bogani G, Serati M, Bolis P. Transumbilical versus transvaginal retrieval of surgical specimens at laparoscopy: a randomized trial. Am J Obstet Gynecol. 2012 Aug;207(2):112.e1-6. doi: 10.1016/j.ajog.2012.05.016. Epub 2012 May 23. PMID 22704765
- [Background] Cohen SL, Clark NV, Ajao MO, Brown DN, Gargiulo AR, Gu X, Einarsson JI. Prospective Evaluation of Manual Morcellation Techniques: Minilaparotomy versus Vaginal Approach. J Minim Invasive Gynecol. 2019 May-Jun;26(4):702-708. doi: 10.1016/j.jmig.2018.07.020. Epub 2018 Aug 1. PMID 30075302